CLINICAL TRIAL: NCT04107272
Title: Evaluating the Use of Repetitive Transcranial Magnetic Stimulation in Cancer Patients With Chemotherapy-Induced Peripheral Neuropathy: A Randomized Feasibility Study
Brief Title: Use of Repetitive Transcranial Magnetic Stimulation in Cancer Patients With Chemotherapy-Induced Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20201116005
Record Dates: First submitted 2019-09-18; First posted 2019-09-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy-induced Peripheral Neuropathy; Repetitive transcranial magnetic stimulation; Pain; Feasibility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Real rTMS
  Interventions: Device: Real repetitive transcranial magnetic stimulation
- Control group (Sham Comparator): Sham rTMS
  Interventions: Device: Sham repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Real repetitive transcranial magnetic stimulation — The real rTMS will be delivered over M1 (hand representation) of dual hemispheres with 10 trains of 10 Hz pulses for 10 seconds, with a total of 1,000 pulses per hemisphere. The real rTMS intensity will be set as 80% resting motor threshold and the interval between each train of pulses will be set as 50 seconds. The real rTMS will be delivered as daily session for five consecutive days, followed by two fortnightly maintenance sessions during the follow-up period after the completion of five daily sessions. The real rTMS will be delivered by designated physical therapists using "figure-of-8" shaped coil.
  Arms: Experimental group
Device: Sham repetitive transcranial magnetic stimulation — The sham rTMS of this study will be delivered with the same active coil angled 90-degree way from the scalp. The intensity of sham rTMS will be set at lowest stimulator output that can generate similar noise to the real rTMS. The sham rTMS will be delivered in the same manner and duration with real rTMS.
  Arms: Control group

SUMMARY:
The study aims to evaluate the feasibility of a repetitive transcranial magnetic simulation (rTMS) protocol developed for managing pain and other related symptoms associated with chemotherapy-induced peripheral neuropathy in cancer patients.

DETAILED DESCRIPTION:
A total of 60 cancer patients who are aged 18 years or above and have persistent peripheral neuropathy for at least 3 months after completion of oxaliplatin-, paclitaxel-, or docetaxel-based chemotherapy will be recruited. After randomization, the experimental group (n = 30) will receive high-frequency rTMS, while the control group (n = 30) will receive sham rTMS. The rTMS will be delivered over M1 (hand representation) of dual hemispheres with 10 trains of 10 Hz pulses for 10 seconds, with a total of 1,000 pulses per hemisphere. The rTMS intensity will be set as 80% resting motor threshold and the interval between each train of pulses will be set as 50 seconds. The rTMS will be delivered as daily session for five consecutive days, followed by two fortnightly maintenance sessions during the follow-up period after the completion of five daily sessions. The rTMS will be delivered by designated physical therapists using "figure-of-8" shaped coil connected to an electromagnetic stimulator in the rehabilitation therapy room of the study hospitals in mainland China.

The research outcomes are feasibility (1. recruitment: i.e. the length of time spent on recruiting participants, the mean number of participants been recruited each month, and the proportion of eligible patients who are finally recruited in the study; 2. eligibility: the proportion of screened patients meeting the inclusion criteria; 3. retention and attrition rates: the proportion of recruited participants who complete the study or who drop out from the study with or without any reason; and 4. appropriateness of clinical outcome measures: the proportion of incomplete questionnaires and neurological tests, as well as the characteristics of the missing data.), acceptability (Chinese version of the Patients' Global Impression of Change [PGIC] scale), safety, and trend of improvement in pain, other related symptoms, and quality of life by rTMS in cancer patients with CIPN.

ELIGIBILITY:
Inclusion Criteria:

* have completed oxaliplatin-, paclitaxel-, or docetaxel-based chemotherapy for at least 3 months;
* complain of persistent symptoms associated with CIPN such as numbness, tingling, burning, or pain with scores ≥ 4 on a numerical rating scale for average daily intensity (0-10, with 10 being the worst) and/or determined as grade 2 or higher CIPN by oncologist according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 (2017);
* with decreased vibration and/or pinprick sensations according to neurological test (provided by the doctoral researcher when patients was referred by their oncologists);
* have a Karnofsky Performance Score ≥ 70;
* can travel to the research hospitals for receiving the study intervention.

Exclusion Criteria:

* having brain tumor or brain metastasis;
* having pregnancy;
* having implanted medical devices;
* having history of epilepsy, brain lesion, head trauma, neurosurgical procedures, or intracranial hypertension;
* having a diagnosis of psychiatric disorder (e.g. bipolar, ongoing major depression, or schizophrenia) and/or treating with antipsychotic drugs;
* having preexisting peripheral neuropathy before initiation of chemotherapy; g) withdrawing from alcohol or sedative medications;
* having a life expectancy less than six months;
* treating with naloxone, which can block analgesic effect of rTMS over M1;
* previously treated with rTMS. Patients receiving any other treatment for CIPN may not be excluded, but they will be required not to change the type and dosage of the current treatments. Furthermore, such information will be collected as baseline clinical data and will be treated as confounding factors during data analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Eligibility rate | Through study completion, an average of 1 year.
  The proportion of screened patients meeting the inclusion criteria.
Recruitment time | Through study completion, an average of 1 year.
  The mean number of participants been recruited each month.
Recruitment rate | Through study completion, an average of 1 year.
  The proportion of eligible patients who are finally recruited in the study.
Retention/attrition rate | Through study completion, an average of 1 year.
  The proportion of recruited participants who complete the study or who drop out from the study with or without any reason.
Appropriateness of clinical outcome measures | Through study completion, an average of 1 year.
  The proportion of incomplete questionnaires and neurological tests.
Participants' perceived effectiveness | Baseline up to 5 weeks
  In this study, affective attitude and perceived effectiveness will be measured by using the Chinese version of the Patient Global Impression of Change (PGIC) scale, a single-item 7-point numerical rating scale from 1 to 7 demonstrating participants' subjective perception of improvement and satisfaction after receiving the intervention (Hurst & Bolton, 2004). The PGIC scale has been recommended by the rTMS research guideline for pain (Klein et al., 2015).

SECONDARY OUTCOMES:
Pain perception | Baseline up to 5 weeks
  The Chinese version of the Brief Pain Inventory (BPI) will be used to assess pain associated with CIPN. This instrument was developed and validated by Wang et al. (2009) for measuring severity (four scales) and interference (seven scales) of pain in cancer patients, which demonstrated good internal consistencies of both domains (Cronbach's α were 0.894 and 0.915, respectively).
Neuropathic symptoms and signs | Baseline up to 5 weeks
  Total Neuropathy Score-nurse© (TNSn©) is a validated instrument to evaluate symptoms and signs associated with CIPN based on both patient-reported and clinician-assessed data including three symptom questions (distribution areas of numbness, tingling/paresthesias, and neuropathic pain) and testing of vibration and pinprick; each of the symptoms and signs is scored from 0 to 4, with higher score indicating worse condition (Smith, Cohen, Pett & Beck, 2010).
Miscellaneous symptoms associated with CIPN | Baseline up to 5 weeks
  The Chinese version of Edmonton Symptom Assessment System (C-ESAS) validated by Dong et al. (2015) will be used to explore whether the intervention would bring any change in the concurrently reported symptoms among cancer patients including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, sleep, well-being, shortness of breath, and potential miscellaneous symptoms that are not listed. Cronbach's α of the C-ESAS was 0.72, indicating an acceptable internal consistency.
Health-related quality of life | Baseline up to 5 weeks
  Functional Assessment of Cancer Therapy-General questionnaire (FACT-G), a widely used self-reported questionnaire measuring health-related quality-of-life (QoL) in cancer patients, will be used in this study. Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale (FACT/GOG-Ntx) will be used to measure the participants' CIPN specific quality of life in this study. It is an 11-item tool added to the FACT measurement system for assessing cancer patients' symptoms and interference induced by neuropathy, which includes sensory, motor, and hearing problems, as well as dysfunctions associated with neuropathy. Good psychometrical properties of the FACT/GOG-Ntx have been demonstrated.
Adverse Effects | Baseline up to 5 weeks
  To determine the safety of rTMS in this population, participants will be asked to report any adverse effect occur during the study. The adverse effects, including the type, occurrence, and duration, will be recorded using a standard form. According to the guidelines (Klein et al., 2015; Rossi et al., 2009), the potential adverse effects associated with rTMS are transient seizures, headaches, transient hearing changes, local pain, neck pain, toothache, and paresthesia. These potential adverse effects will be listed in the standard form, and will be filled out by the designated therapists based on their observation and the participants' self-report after each treatment session. If any adverse effect occurs but is not listed in the form, the therapist will record the condition in the "Other" column.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University